CLINICAL TRIAL: NCT06183749
Title: Predictors of Mortality in Patients With Traumatic Brain Injury in the Tertiary Intensive Care Unit
Brief Title: Predictors of Mortality in Traumatic Brain Injury Patients in Intensive Care Unit
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Senay Goksu, SPECIALIST, MD,, Umraniye Education and Research Hospital
Other Study IDs: trauma
Record Dates: First submitted 2023-12-12; First posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Brain Injuries, Traumatic
Keywords: brain injuries, traumatic, mortality prediction
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries | interventions — Hospitalization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1general body trauma (Group 1): Diagnosed as traumatic brain injury due to general body trauma neurosurgery in the emergency department and hospitalized for more than 24 hours in the 3rd stage Anesthesiology and Reanimation unit and those who have been in intensive care within the past two years.
  Interventions: Other: hospitalisation for more than 24 hours in the 3rd stage Anesthesiology and Reanimation unit
- isolated head trauma (Group 2).: diagnosed as traumatic brain injury due isolated head trauma neurosurgery in the emergency department and hospitalized for more than 24 hours in the 3rd stage Anesthesiology and Reanimation unit and those who have been in intensive care within the past two years.
  Interventions: Other: hospitalisation for more than 24 hours in the 3rd stage Anesthesiology and Reanimation unit

INTERVENTIONS:
Other: hospitalisation for more than 24 hours in the 3rd stage Anesthesiology and Reanimation unit — diagnosed as traumatic brain injury by neurosurgery in the emergency department and hospitalized for more than 24 hours in the 3rd stage Anesthesiology and Reanimation unit and receivied appropriate necessary treatment

SUMMARY:
The primary outcome of this study was to identify mortality predictors/risk factors affecting mortality and secondary outcome was to determine the distribution of brain injury types and other parameters according to type of trauma in patients with TBI treated in anesthesia-reanimation tertiary ICU.

DETAILED DESCRIPTION:
Patients with traumatic brain injury (TBI), especially severe cases are referred to neurotrauma centers where they are managed in neurosurgery intensive care units (ICU) or anesthesia-reanimation intensive care units as in Turkey. Such patients comprise a significant portion of patients managed in ICU with high rates of mortality and morbidity even with the best medical and neurosurgical care. It is crucial to identify the factors that contribute to mortality for TBI as it has a high incidence rate with significant mortality and morbidity.The aim of this study was to identify mortality predictors/risk factors affecting mortality and was to assess the distribution of brain injury in patients with TBI in anesthesia-reanimation ICU.

After receiving approval from the institutional Ethics Committee, we retrospectively identified patients over the age of 18 who were diagnosed with TBI by neurosurgery in the emergency department and were hospitalized in the 3rd stage Anesthesiology and Reanimation-ICU for more than 24 hours, within the last two-years period, using hospital computer records. They were then included in our studyThe patients were evaluated in 2 groups according to etiology as head trauma accompanied by general body trauma (Group 1) and isolated head trauma (Group 2).

Types of brain injury/hemorrhage due to head trauma were determined as intracerebral hemorrhage (ICH), subdural hematoma (SDH), epidural hematoma (EDH), traumatik subarachnoid hemorrhage (tSAH), cerebral contusion-diffuse axonal injury (DAI), and hemorrhages in which two or more of these conditions were combined (MIX).

Parameters included; age, sex, GCS at admission, APACHE II score, estimated mortality, actual mortality, type of brain injury, presence or absence of surgical intervention, presence or absence of skull fracture, length of ICU stay, duration of intubation, presence or absence of sedation, presence or absence of tracheotomy and outcome of disease. All data regarding above-mentioned parameters were extracted from patient files and electronic database.

It was aimed to assess relationship between mortality and parameters such as age, sex, surgical intervention, type of brain injury, duration of intubation, duration in ICU, GCS score and APACHE II scores, skull fracture in cases with TBI as primary outcome, it was also aimed to determine the distribution of etiology and these parameters over the TBI patients as secondary outcome.

As surgical intervention, operations with indications of bleeding control and/or control of intracranial pressure performed by neurosurgery department were taken into consideration for analysis.

In all patients, diagnosis was made based on CT scan and/or MR imaging study obtained at arrival to emergency department as a part of emergency protocol.

ELIGIBILITY:
Inclusion Criteria:

* patients over the age of 18,
* diagnosed as traumatic brain injury by neurosurgery in the emergency department .hospitalized for more than 24 hours in the 3rd stage Anesthesiology and Reanimation unit

Exclusion Criteria:

Failure to obtain institutional Ethics Committee approval Failure to obtain patients records

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients over the age of 18, diagnosed as traumatic brain injury by neurosurgery in the emergency department and hospitalized for more than 24 hours in the 3rd stage Anesthesiology and Reanimation unit
Sampling Method: Non-Probability Sample
Enrollment: 194 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
mortality predictor | through study completion, an average of 2 months
  Identification of those that are associated with mortality among the parameters examined

IPD SHARING:
Plan to Share IPD: No